CLINICAL TRIAL: NCT03066635
Title: Botulinum Toxin Type A Block of the Otic Ganglion in Chronic Cluster Headache: Safety Issues
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTOBLOCKCH2016; 2016-004213-28 (EudraCT Number)
Record Dates: First submitted 2017-02-13; First posted 2017-02-28 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Cluster Headache
Keywords: Nerve block; Ganglia, Parasympathetic; Botulinum Toxins, Type A; Injection
MeSH Terms: conditions — Cluster Headache; Ganglion Cysts | interventions — Botulinum Toxins, Type A; Idoxuridine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum Toxin 25 IU (Experimental): 5 patients will be injected with 25 IU of Botulinum Toxin Type A towards the otic ganglion in the symptomatic side (ipsilateral to the pain)
  Interventions: Drug: Botulinum Toxin Type A 25 IU
- Botulinum Toxin 12.5 IU (Experimental): 5 patients will be injected with 12.5 IU of Botulinum Toxin Type A towards the otic ganglion in the symptomatic side (ipsilateral to the pain)
  Interventions: Drug: Botulinum Toxin Type A 12.5 IU

INTERVENTIONS:
Drug: Botulinum Toxin Type A 25 IU — injection with 25 IU botulinum toxin towards the otic ganglion (symptomatic side) using image-guided navigation and the MultiGuide device
  Other Names: Botox; BTA; Allergan
  Arms: Botulinum Toxin 25 IU
Drug: Botulinum Toxin Type A 12.5 IU — injection with 12.5 IU botulinum toxin towards the otic ganglion (symptomatic side) using image-guided navigation and the MultiGuide device
  Other Names: Botox; BTA; Allergan
  Arms: Botulinum Toxin 12.5 IU

SUMMARY:
Cluster headache (CH) is the most common of the trigeminal autonomic cephalalgias and one of the most severe pains known to man, having a large impact on the sufferer's quality of life. A parasympathetic dysfunction in CH has been suggested. The sphenopalatine ganglion has been a target for treatment of primary headache disorders for more than a century but there are several anatomic and physiologic studies that suggest that another cranial parasympathetic ganglion, the otic ganglion (OG), might be also relevant in CH. In this study OG will be blocked with botulinum toxin type A in a pilot study in 10 patients with chronic cluster headache. Recruitment of patients will be solely in Norway. There is no data available to determine the correct dosage of botulinum toxin. A similar neural structure that has been blocked with botulinum toxin in humans is the sphenopalatine ganglion. The investigators injected 10 patients suffering from intractable chronic cluster headache with botulinum toxin in the sphenopalatine ganglion. 5 patients were given 25 IU and 5 patients were given 50 IU. Even though the number of treated patients is low, there did not appear to be differences in the adverse events profile between those who received 25 Iu and those who received 50 IU. The investigators also previously injected 25 IU botulinum toxin towards the sphenopalatine ganglion bilaterally (i.e. 25 IU in each side) in 10 patients suffering from intractable chronic migraine. Doses of up to 25 IU have been injected in structures adjacent to the otic ganglion, for instance in dystonia towards the lateral pterygoid muscle. Thus it was decided for this study on injection towards the otic ganglion, to explore the safety of 12.5 and 25 IU of botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Fulfilling International Classification of Headache Disorders (ICHD) -3 Beta criteria for chronic cluster headache
* Mean attack frequency of four attacks per week or more
* Agreeing to refrain from starting new prophylactic cluster headache medication, including steroids, or any other therapy aimed at cluster headache, and agreeing to maintain existing prophylactic cluster headache medication from 4 weeks before entering the baseline period throughout the duration of the study
* Intractable cluster headache, i.e. unsatisfactory effect, intolerable side effects or contraindication of at least 2 of the following medications: Verapamil, Lithium, Suboccipital steroid injection,
* Able to distinguish between cluster headache attacks and other types of headache.

Exclusion Criteria:

* Modification or addition of any prophylactic drug dose used against cluster headache in the last 4 weeks before inclusion of during the trial
* Use of antipsychotic medication in the last 4 weeks before inclusion
* Concomitant significant heart or lung disease
* Systemic or local conditions which can increase the risk of the procedure
* Psychiatric or psychological conditions interfering with the participation in the study
* Pregnancy
* Breast feeding
* Inadequate use of contraceptives
* Opioid overuse
* Abuse of drugs including alcohol
* Anatomical variants which might impede the study treatment
* Known hypersensitivity to botulinum toxin type A or any of the excipients found in Botox
* Current treatment with drugs that interact with botulinum toxin: aminoglycosides, spectinomycin, neuromuscular blockers, both depolarizing agents (such as succinylcholine) or non-depolarizing agents (tubocurarine derivates), lincosamides, polymyxins, quinidine, magnesium sulfate or anticholinesterases.
* Previous cerebral ischemic infarction
* Not able to take magnetic resonance imaging (MRI)
* Previous destructive surgery of interventional procedures involving the C2 and C3 roots (vertebrae), sphenopalatine ganglion, any extracranial nerve, trigeminal nerve, or deep brain stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AE) | for the follow-up period of 6 months
  All adverse events will be registered. The likelihood of a relationship between the AE and the pharmacological substance or the procedure will be evaluated. Data will be collected from the headache diary (free text) and open questions at the office follow up visits.

SECONDARY OUTCOMES:
Number of cluster headache attacks per week | for the follow-up period of 6 months
  Number of cluster headache attacks per week
Duration of cluster headache attacks | for the follow-up period of 6 months
  Duration of cluster headache attacks
Days without cluster headache attacks | for the follow-up period of 6 months
  number of days without cluster headache attacks
Headache intensity on a 0-5 scale | for the follow-up period of 6 months
  The headache intensity is registered in the headache diary using a scale from 0-5
Mean intensity per attack | for the follow-up period of 6 months
  The headache intensity is registered in the headache diary using a scale from 0-5
Mean number of attacks with intensity grade 4-5 | for the follow-up period of 6 months
  Mean number of attacks with intensity grade 4-5
Functional level | for the follow-up period of 6 months
  The functional level will be assessed by the WHO Performance Status
Triptan use per 4 weeks | for the follow-up period of 6 months
  Triptan use per 4 weeks during the whole duration of the study
Number of analgesic doses per 4 weeks | for the follow-up period of 6 months
  the number of analgesic doses per 4 weeks during the whole duration of the study
Absenteeism due to cluster headache | for the follow-up period of 6 months
  Absenteeism due to cluster headache as assessed by the headache diary
disability | for the follow-up period of 6 months
  as assessed by a qualitative questionnaire (HIT-6)
Occurrence of autonomic symptoms | for the follow-up period of 6 months
  assessed on Cranial Autonomic Parasympathetic Symptoms (CAPS) scale

CONTACTS AND LOCATIONS:
Overall Officials: Lars Jacob Stovner, prof MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Crespi J, Bratbak D, Dodick DW, Matharu M, Solheim O, Gulati S, Berntsen EM, Tronvik E. Open-Label, Multi-Dose, Pilot Safety Study of Injection of OnabotulinumtoxinA Toward the Otic Ganglion for the Treatment of Intractable Chronic Cluster Headache. Headache. 2020 Sep;60(8):1632-1643. doi: 10.1111/head.13889. Epub 2020 Jun 25. PMID 32583902